CLINICAL TRIAL: NCT03736278
Title: Retrospective Analysis of Tuberculosis in Rheumatic Diseases for Epidemiology, Risk Factors, Disease Presentation, Complications, Treatment, and Prognosis
Brief Title: Characteristics of Tuberculosis Infection in Rheumatic Disease
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201805069RIND
Record Dates: First submitted 2018-11-04; First posted 2018-11-09 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2018-06

CONDITIONS: Tuberculosis; Autoimmune Diseases
MeSH Terms: conditions — Tuberculosis; Autoimmune Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — We group the patients according to the outcome (survival vs mortality)

SUMMARY:
A retrospective study evaluating the characteristics of tuberculosis infection in patients of rheumatic disease.

ELIGIBILITY:
Inclusion Criteria:

* The patients with International Classification of Diseases (ICD) codes of rheumatic diseases during 2006-2017
* Definite evidence of tuberculosis infection

Exclusion Criteria:

* HIV, malignancy, not follow-up rheumatic disease in National Taiwan University Hospital, younger than 20-year-old, refusing attend research

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients of rheumatic disease
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-11-10 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2019-09-24 (Actual)

PRIMARY OUTCOMES:
Mortality | approximately 6 months
  Death of any cause (The definition of TB mortality from WHO is death of any cause during TB treatment.)

CONTACTS AND LOCATIONS:
Overall Officials: Chiao-Feng Cheng, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided